CLINICAL TRIAL: NCT06890143
Title: The Efficacy and Safety of Dapagliflozin in the Treatment of Hereditary Kidney Disease With Proteinuria in Children: a Prospective, Randomized Crossover Trial
Brief Title: The Efficacy and Safety of Dapagliflozin in the Treatment of Hereditary Kidney Disease With Proteinuria in Children
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Guangzhou Women and Children's Medical Center (Other); Maternal and Child Health Hospital of Guangxi Zhuang Autonomous Region (Other); Shandong Provincial Hospital (Other Government); The First Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other); Wuhan Children's Hospital (Other); Xuzhou Children Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Kunming Children's Hospital (Other); The Children's Hospital of Zhejiang University School of Medicine (Other); Children's Hospital of Nanjing Medical University (Other); Zhengzhou Children's Hospital, China (Other); Xiamen Women's and Children's Hospital (Unknown); Guiyang Maternity and Child Health Care Hospital (Other); Maternal and Child Health Care Hospital of Hainan Province (Other); Children's Hospital of The Capital Institute of Pediatrics (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Xian Children's Hospital (Other Government); The Second Hospital of Hebei Medical University (Other); Wuxi Women's & Children's Hospital (Other); First People's Hospital of Urumqi (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: DAPA-PedHKD
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Pediatric Hereditary Kidney Diseases
Keywords: hereditary kidney diseases; proteinuria; dapagliflozin; children
MeSH Terms: conditions — Proteinuria

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Dapagliflozin Group (Experimental): ①Dapagliflozin+Standard Treatment for 12 weeks. Dapagliflozin therapy (Farxiga®, 10 mg tablets) is administered orally once daily,with dose adjustment based on body weight.Standard Treatment:standard renin-angiotensin-aldosterone system inhibitor (RAASi) therapy(The dosage will be maintained at the pre-enrollment level throughout the entire treatment period, with no adjustments made during therapy.),This combined therapy will be administered for 12 weeks.
  ② Washout period for 4 weeks Participants should maintain RAASi therapy while discontinuing dapagliflozin.
  ③RAASi monotherapy alone for an additional 12 weeks.
  Interventions: Drug: Dapagliflozin+Standard Treatment for 12 weeks,washout period for 4 weeks，then Standard Treatment alone for12 weeks
- Delayed Dapagliflozin Group (Experimental): ① Standard Treatment for 12 weeks Standard Treatment:Standard renin-angiotensin-aldosterone system inhibitor (RAASi) therapy alone for 12 weeks.(The dosage will be maintained at the pre-enrollment level throughout the entire treatment period, with no adjustments made during therapy.)
  ② Washout period for 4 weeks Participants should maintain RAASi therapy without additional interventions.
  ③ Dapagliflozin+Standard Treatment for 12 weeks Dapagliflozin therapy is administered orally once daily,with dose adjustment based on body weight.This combined therapy will be administered for 12 weeks.
  Interventions: Drug: Standard Treatment alone for 12 weeks ,washout period for 4 weeks ,then Dapagliflozin+Standard Treatment for 12 weeks

INTERVENTIONS:
Drug: Dapagliflozin+Standard Treatment for 12 weeks,washout period for 4 weeks，then Standard Treatment alone for12 weeks — ①Dapagliflozin+Standard Treatment for 12 weeks. Dapagliflozin therapy (Farxiga®, 10 mg tablets) is administered orally once daily,with dose adjustment based on body weight: 5 mg/day for participants ≤30 kg; 5 mg/day initially (first week), then increased to 10 mg/day for participants >30 kg Standard Treatment:standard renin-angiotensin-aldosterone system inhibitor (RAASi) therapy(The dosage will be maintained at the pre-enrollment level throughout the entire treatment period, with no adjustments made during therapy.),This combined therapy will be administered for 12 weeks.
  ② Washout period for 4 weeks Participants should maintenance RAASi therapy while discontinuing dapagliflozin.
  ③Standard Treatment alone for an additional 12 weeks. To ensure compliance, all participants are required to complete a daily medication log.If any adverse events (AEs) occur, appropriate clinical interventions will be promptly implemented
  Arms: Early Dapagliflozin Group
Drug: Standard Treatment alone for 12 weeks ,washout period for 4 weeks ,then Dapagliflozin+Standard Treatment for 12 weeks — ①Standard Treatment for 12 weeks Standard Treatment:Standard renin-angiotensin-aldosterone system inhibitor (RAASi) therapy alone for 12 weeks.(The dosage will be maintained at the pre-enrollment level throughout the entire treatment period, with no adjustments made during therapy.)
  ②Washout period for 4 weeks Participants should maintenance RAASi therapy while discontinuing dapagliflozin.
  ③Dapagliflozin+Standard Treatment for 12 weeks Dapagliflozin therapy (Farxiga®, 10 mg tablets) is administered orally once daily,with dose adjustment based on body weight: 5 mg/day for participants ≤30 kg; 5 mg/day initially (first week), then increased to 10 mg/day for participants >30 kg.This combined therapy will be administered for 12 weeks To ensure compliance, all participants are required to complete a daily medication log.If any adverse events (AEs) occur, appropriate clinical interventions will be promptly implemented
  Arms: Delayed Dapagliflozin Group

SUMMARY:
This study is a multicenter, randomized controlled crossover trial aimed to evaluate the efficacy and safety of dapagliflozin in the treatment of hereditary kidney disease with proteinuria in children

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) poses a significant public health threat to children, with hereditary kidney diseases exhibiting limited therapeutic efficacy in reducing proteinuria. Global studies have demonstrated that dapagliflozin significantly reduces proteinuria in adults with CKD; however, its role in pediatric hereditary kidney diseases lacks strong evidence .This study aims to investigate the efficacy and safety of dapagliflozin in children with proteinuric hereditary kidney diseases.

This is a multicenter, open-label, block-randomized, crossover clinical trial with 1:1 allocation. A total of 44 participants will be enrolled to compare the efficacy and safety of dapagliflozin combined with standard renin-angiotensin-aldosterone system inhibitor (RAASi) therapy versus RAASi therapy alone.

The primary endpoint is the change in 24-hour urinary protein levels from baseline to 12 weeks of treatment. Secondary endpoints include: urinary protein-to-creatinine ratio (UPCR), urinary albumin-to-creatinine ratio (UACR), serum albumin levels, estimated glomerular filtration rate (eGFR), blood pressure changes, and body weight changes.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of hereditary kidney disease (identification of pathogenic genes through molecular genetic testing; for Alport syndrome, molecular diagnosis is not necessarily required if diagnosed based on clinical and pathological findings; for those with a clear family history and a high clinical suspicion of hereditary kidney disease).
* 24 - hour urinary protein level > 0.2 g or urinary protein to creatinine ratio (UPCR) > 0.2 mg/mg.
* Calculate the estimated glomerular filtration rate (eGFR) using the Schwartz formula (36.5 * height in cm / serum creatinine in μmol/L), with eGFR ≥ 60 ml/min/1.73 m².
* Stable use of the basic treatment drug RAASi (including ACEI/ARB) for more than 4 weeks, and no dosage adjustment during the treatment period.
* Willingness to sign the informed consent form.

Exclusion Criteria:Exclusion applies if any of the following criteria are met:

* Treatment with hormones/immunosuppressive agents within the previous 4 weeks.
* Treatment with SGLT2 inhibitors within the previous 4 weeks.
* Comorbid diabetes.
* Uncontrolled urinary tract infection.
* Evidence of urinary tract obstruction such as dysuria.
* Blood pressure below the 5th percentile for the same gender, age, and height.
* Organ transplantation.
* Tumor.
* Presence of any of the following definite evidence of liver disease: ALT/AST reaching 2 times the normal value, hepatic encephalopathy, esophageal varices, or portal shunt surgery.
* Comorbid medical conditions that may affect drug absorption, distribution, metabolism, and excretion, including but not limited to any of the following: active inflammatory bowel disease within the past 6 months, history of major gastrointestinal surgery (such as gastrectomy, gastroenterostomy, intestinal resection), gastrointestinal ulcer, gastrointestinal or rectal bleeding within the past 6 months, pancreatic injury or pancreatitis within the past 6 months.
* Subjects at risk of dehydration or volume depletion, which may affect drug efficacy or safety.
* Participation in other drug trials within the previous 4 weeks.
* Blood loss exceeding 400 ml within the previous 8 weeks.
* Poor past medication compliance or unwillingness to complete the trial.
* Any other medical conditions that may place the patient at a higher risk due to participation in this study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — gender based.
Enrollment: 44 (Estimated)
Dates: Start 2025-03-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes in 24-hour urinary protein excretion from baseline to week 12 | From baseline to week 12
  The change in 24-hour urinary protein excretion from baseline to week 12 of treatment with dapagliflozin combined with RAASi . According to the research protocol, the 24-hour urine of the pediatric patients is collected during the planned follow-up period, and the pyrogallol red method is used for the quantitative test of the protein in the urine.

SECONDARY OUTCOMES:
Changes in urinary protein to creatinine ratio (UPCR) levels from baseline to week 12 | From baseline to week 12
  The change in the urinary protein to creatinine ratio (UPCR) levels from baseline to week 12 of treatment with dapagliflozin combined with RAASi. The pyrogallol red method is used for detecting urinary protein, and the enzymatic method is used for detecting urinary creatinine. UPCR = urinary protein/urinary creatinine (mg/mg).
Changes in urinary albumin to creatinine ratio (UACR) levels from baseline to week 12 | From baseline to week 12
  The change in urinary albumin to creatinine ratio (UACR) levels from baseline to week 12 of treatment with dapagliflozin combined with RAASi. The immunoturbidimetric method is used for detecting urinary albumin, and the enzymatic method is used for detecting urinary creatinine. UACR = urinary albumin/urinary creatinine (mg/g).
Changes in serum albumin levels from baseline to week 12 | From baseline to week 12
  The change in the serum albumin level from baseline to week 12 of treatment with dapagliflozin combined with RAASi. Venous blood is collected, and the test is conducted through the routine biochemical examination in the hospital.
Changes in estimated glomerular filtration rate from baseline to week 12 | From baseline to week 12
  The change in the estimated glomerular filtration rate (eGFR) from baseline to week 12 of treatment with dapagliflozin combined with RAASi. Venous blood is collected, and the serum creatinine level is detected through the routine biochemical examination in the hospital. The eGFR is calculated according to the Schwartz formula (36.5 * height in cm / serum creatinine in μmol/L).
Changes in blood pressure from baseline to week 12 | From baseline to week 12
  The change in both systolic and diastolic blood pressure from baseline to week 12 of treatment with dapagliflozin combined with RAASi. The measurement is taken after the pediatric patient sits quietly for 5 minutes.
Changes in weight from baseline to week 12 | From baseline to week 12
  The change in body weight from baseline to week 12 of treatment with dapagliflozin combined with RAASi. The measurement is taken using a calibrated weighing scale.

CONTACTS AND LOCATIONS:
Overall Officials: YIHUI ZHAI, Study Director — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Chinese Preventive Medicine Association for Kidney Disease. [Guidelines for the early evaluation and management of chronic kidney disease in China]. Zhonghua Nei Ke Za Zhi. 2023 Aug 1;62(8):902-930. doi: 10.3760/cma.j.cn112138-20221013-00755. Chinese. PMID 37528029
- [Background] The Expert Group of Chinese Expert Consensus on the Clinical Application of Sodium-glucose Cotransporter 2 Inhibitors in Patients with Chronic Kidney Disease. Chinese expert consensus on the clinical application of sodium-glucose cotransporter 2 inhibitors in patients with chronic kidney disease. Chin Med J (Engl). 2024 Jun 5;137(11):1264-1266. doi: 10.1097/CM9.0000000000003145. Epub 2024 May 13. No abstract available. PMID 38738698
- [Background] O'Hara DV, Lam CSP, McMurray JJV, Yi TW, Hocking S, Dawson J, Raichand S, Januszewski AS, Jardine MJ. Applications of SGLT2 inhibitors beyond glycaemic control. Nat Rev Nephrol. 2024 Aug;20(8):513-529. doi: 10.1038/s41581-024-00836-y. Epub 2024 Apr 26. PMID 38671190
- [Background] Koppe L, Fouque D. The Role for Protein Restriction in Addition to Renin-Angiotensin-Aldosterone System Inhibitors in the Management of CKD. Am J Kidney Dis. 2019 Feb;73(2):248-257. doi: 10.1053/j.ajkd.2018.06.016. Epub 2018 Aug 24. PMID 30149957
- [Background] Herrington WG, Preiss D, Haynes R, von Eynatten M, Staplin N, Hauske SJ, George JT, Green JB, Landray MJ, Baigent C, Wanner C. The potential for improving cardio-renal outcomes by sodium-glucose co-transporter-2 inhibition in people with chronic kidney disease: a rationale for the EMPA-KIDNEY study. Clin Kidney J. 2018 Dec;11(6):749-761. doi: 10.1093/ckj/sfy090. Epub 2018 Oct 25. PMID 30524708
- [Background] Cherney DZI, Dekkers CCJ, Barbour SJ, Cattran D, Abdul Gafor AH, Greasley PJ, Laverman GD, Lim SK, Di Tanna GL, Reich HN, Vervloet MG, Wong MG, Gansevoort RT, Heerspink HJL; DIAMOND investigators. Effects of the SGLT2 inhibitor dapagliflozin on proteinuria in non-diabetic patients with chronic kidney disease (DIAMOND): a randomised, double-blind, crossover trial. Lancet Diabetes Endocrinol. 2020 Jul;8(7):582-593. doi: 10.1016/S2213-8587(20)30162-5. PMID 32559474
- [Background] Heerspink HJL, Cherney D, Postmus D, Stefansson BV, Chertow GM, Dwyer JP, Greene T, Kosiborod M, Langkilde AM, McMurray JJV, Correa-Rotter R, Rossing P, Sjostrom CD, Toto RD, Wheeler DC; DAPA-CKD Trial Committees and Investigators. A pre-specified analysis of the Dapagliflozin and Prevention of Adverse Outcomes in Chronic Kidney Disease (DAPA-CKD) randomized controlled trial on the incidence of abrupt declines in kidney function. Kidney Int. 2022 Jan;101(1):174-184. doi: 10.1016/j.kint.2021.09.005. Epub 2021 Sep 22. PMID 34560136
- [Result] Scheen AJ. Sodium-glucose cotransporter type 2 inhibitors for the treatment of type 2 diabetes mellitus. Nat Rev Endocrinol. 2020 Oct;16(10):556-577. doi: 10.1038/s41574-020-0392-2. Epub 2020 Aug 27. PMID 32855502
- [Result] Ravani P, Rossi R, Bonanni A, Quinn RR, Sica F, Bodria M, Pasini A, Montini G, Edefonti A, Belingheri M, De Giovanni D, Barbano G, Degl'Innocenti L, Scolari F, Murer L, Reiser J, Fornoni A, Ghiggeri GM. Rituximab in Children with Steroid-Dependent Nephrotic Syndrome: A Multicenter, Open-Label, Noninferiority, Randomized Controlled Trial. J Am Soc Nephrol. 2015 Sep;26(9):2259-66. doi: 10.1681/ASN.2014080799. Epub 2015 Jan 15. PMID 25592855
- [Result] Heerspink HJL, Jongs N, Chertow GM, Langkilde AM, McMurray JJV, Correa-Rotter R, Rossing P, Sjostrom CD, Stefansson BV, Toto RD, Wheeler DC, Greene T; DAPA-CKD Trial Committees and Investigators. Effect of dapagliflozin on the rate of decline in kidney function in patients with chronic kidney disease with and without type 2 diabetes: a prespecified analysis from the DAPA-CKD trial. Lancet Diabetes Endocrinol. 2021 Nov;9(11):743-754. doi: 10.1016/S2213-8587(21)00242-4. Epub 2021 Oct 4. PMID 34619108
- [Result] Waijer SW, Vart P, Cherney DZI, Chertow GM, Jongs N, Langkilde AM, Mann JFE, Mosenzon O, McMurray JJV, Rossing P, Correa-Rotter R, Stefansson BV, Toto RD, Wheeler DC, Heerspink HJL. Effect of dapagliflozin on kidney and cardiovascular outcomes by baseline KDIGO risk categories: a post hoc analysis of the DAPA-CKD trial. Diabetologia. 2022 Jul;65(7):1085-1097. doi: 10.1007/s00125-022-05694-6. Epub 2022 Apr 21. PMID 35445820
- [Result] Jongs N, Greene T, Chertow GM, McMurray JJV, Langkilde AM, Correa-Rotter R, Rossing P, Sjostrom CD, Stefansson BV, Toto RD, Wheeler DC, Heerspink HJL; DAPA-CKD Trial Committees and Investigators. Effect of dapagliflozin on urinary albumin excretion in patients with chronic kidney disease with and without type 2 diabetes: a prespecified analysis from the DAPA-CKD trial. Lancet Diabetes Endocrinol. 2021 Nov;9(11):755-766. doi: 10.1016/S2213-8587(21)00243-6. Epub 2021 Oct 4. PMID 34619106
- [Result] HEERSPINK H J L, STEFáNSSON B V, CORREA-ROTTER R, et al. Dapagliflozin in Patients with Chronic Kidney Disease
- [Result] Heerspink HJL, Stefansson BV, Chertow GM, Correa-Rotter R, Greene T, Hou FF, Lindberg M, McMurray J, Rossing P, Toto R, Langkilde AM, Wheeler DC; DAPA-CKD Investigators. Rationale and protocol of the Dapagliflozin And Prevention of Adverse outcomes in Chronic Kidney Disease (DAPA-CKD) randomized controlled trial. Nephrol Dial Transplant. 2020 Feb 1;35(2):274-282. doi: 10.1093/ndt/gfz290. PMID 32030417
- [Result] Rajasekeran H, Reich HN, Hladunewich MA, Cattran D, Lovshin JA, Lytvyn Y, Bjornstad P, Lai V, Tse J, Cham L, Majumder S, Bowskill BB, Kabir MG, Advani SL, Gibson IW, Sood MM, Advani A, Cherney DZI. Dapagliflozin in focal segmental glomerulosclerosis: a combined human-rodent pilot study. Am J Physiol Renal Physiol. 2018 Mar 1;314(3):F412-F422. doi: 10.1152/ajprenal.00445.2017. Epub 2017 Nov 15. PMID 29141939
- [Result] Perkovic V, de Zeeuw D, Mahaffey KW, Fulcher G, Erondu N, Shaw W, Barrett TD, Weidner-Wells M, Deng H, Matthews DR, Neal B. Canagliflozin and renal outcomes in type 2 diabetes: results from the CANVAS Program randomised clinical trials. Lancet Diabetes Endocrinol. 2018 Sep;6(9):691-704. doi: 10.1016/S2213-8587(18)30141-4. Epub 2018 Jun 21. PMID 29937267
- [Result] Kadowaki T, Nangaku M, Hantel S, Okamura T, von Eynatten M, Wanner C, Koitka-Weber A. Empagliflozin and kidney outcomes in Asian patients with type 2 diabetes and established cardiovascular disease: Results from the EMPA-REG OUTCOME(R) trial. J Diabetes Investig. 2019 May;10(3):760-770. doi: 10.1111/jdi.12971. Epub 2019 Jan 7. PMID 30412655
- [Result] Jardine MJ, Mahaffey KW, Neal B, Agarwal R, Bakris GL, Brenner BM, Bull S, Cannon CP, Charytan DM, de Zeeuw D, Edwards R, Greene T, Heerspink HJL, Levin A, Pollock C, Wheeler DC, Xie J, Zhang H, Zinman B, Desai M, Perkovic V; CREDENCE study investigators. The Canagliflozin and Renal Endpoints in Diabetes with Established Nephropathy Clinical Evaluation (CREDENCE) Study Rationale, Design, and Baseline Characteristics. Am J Nephrol. 2017 Dec 13;46(6):462-472. doi: 10.1159/000484633. Online ahead of print. PMID 29253846
- [Result] Heerspink HJ, Desai M, Jardine M, Balis D, Meininger G, Perkovic V. Canagliflozin Slows Progression of Renal Function Decline Independently of Glycemic Effects. J Am Soc Nephrol. 2017 Jan;28(1):368-375. doi: 10.1681/ASN.2016030278. Epub 2016 Aug 18. PMID 27539604
- [Result] Tirucherai GS, LaCreta F, Ismat FA, Tang W, Boulton DW. Pharmacokinetics and pharmacodynamics of dapagliflozin in children and adolescents with type 2 diabetes mellitus. Diabetes Obes Metab. 2016 Jul;18(7):678-84. doi: 10.1111/dom.12638. PMID 27291448
- [Result] Dekkers CCJ, Gansevoort RT, Heerspink HJL. New Diabetes Therapies and Diabetic Kidney Disease Progression: the Role of SGLT-2 Inhibitors. Curr Diab Rep. 2018 Mar 27;18(5):27. doi: 10.1007/s11892-018-0992-6. PMID 29589183
- [Result] Vallon V, Thomson SC. Targeting renal glucose reabsorption to treat hyperglycaemia: the pleiotropic effects of SGLT2 inhibition. Diabetologia. 2017 Feb;60(2):215-225. doi: 10.1007/s00125-016-4157-3. Epub 2016 Nov 22. PMID 27878313
- [Result] Petrovic D, Stojimirovic B. Proteinuria as a risk factor for the progression of chronic renal disease. Vojnosanit Pregl. 2008 Jul;65(7):552-8. doi: 10.2298/vsp0807552p. No abstract available. PMID 18700466
- [Result] Jafar TH, Stark PC, Schmid CH, Landa M, Maschio G, Marcantoni C, de Jong PE, de Zeeuw D, Shahinfar S, Ruggenenti P, Remuzzi G, Levey AS; AIPRD Study Group. Angiotensin-Converting Enzymne Inhibition and Progression of Renal Disease. Proteinuria as a modifiable risk factor for the progression of non-diabetic renal disease. Kidney Int. 2001 Sep;60(3):1131-40. doi: 10.1046/j.1523-1755.2001.0600031131.x. PMID 11532109
- [Result] Leung AK, Wong AH, Barg SS. Proteinuria in Children: Evaluation and Differential Diagnosis. Am Fam Physician. 2017 Feb 15;95(4):248-254. PMID 28290633
- [Result] Sumida K, Molnar MZ, Potukuchi PK, George K, Thomas F, Lu JL, Yamagata K, Kalantar-Zadeh K, Kovesdy CP. Changes in Albuminuria and Subsequent Risk of Incident Kidney Disease. Clin J Am Soc Nephrol. 2017 Dec 7;12(12):1941-1949. doi: 10.2215/CJN.02720317. Epub 2017 Sep 11. PMID 28893924
- [Result] Romagnani P, Remuzzi G, Glassock R, Levin A, Jager KJ, Tonelli M, Massy Z, Wanner C, Anders HJ. Chronic kidney disease. Nat Rev Dis Primers. 2017 Nov 23;3:17088. doi: 10.1038/nrdp.2017.88. PMID 29168475
- [Result] Yang CW, Harris DCH, Luyckx VA, Nangaku M, Hou FF, Garcia Garcia G, Abu-Aisha H, Niang A, Sola L, Bunnag S, Eiam-Ong S, Tungsanga K, Richards M, Richards N, Goh BL, Dreyer G, Evans R, Mzingajira H, Twahir A, McCulloch MI, Ahn C, Osafo C, Hsu HH, Barnieh L, Donner JA, Tonelli M. Global case studies for chronic kidney disease/end-stage kidney disease care. Kidney Int Suppl (2011). 2020 Mar;10(1):e24-e48. doi: 10.1016/j.kisu.2019.11.010. Epub 2020 Feb 19. PMID 32149007
- [Result] Zhang L, Wang F, Wang L, Wang W, Liu B, Liu J, Chen M, He Q, Liao Y, Yu X, Chen N, Zhang JE, Hu Z, Liu F, Hong D, Ma L, Liu H, Zhou X, Chen J, Pan L, Chen W, Wang W, Li X, Wang H. Prevalence of chronic kidney disease in China: a cross-sectional survey. Lancet. 2012 Mar 3;379(9818):815-22. doi: 10.1016/S0140-6736(12)60033-6. PMID 22386035
- [Derived] Zhang W, Dou Y, Liu J, Liu T, Yan W, Shen Q, Xu H, Zhai Y. Effects and safety of dapagliflozin in paediatric hereditary kidney disease: protocol for a multicentric, prospective, open and randomised crossover study (DAPA-PedHKD). BMJ Open. 2025 Dec 14;15(12):e109833. doi: 10.1136/bmjopen-2025-109833. PMID 41397763